CLINICAL TRIAL: NCT06229886
Title: Effect of Positive End-Expiratory Pressure on Tricuspid Regurgitant Jet Velocity in Pediatric Patients on Invasive Mechanical Ventilation
Brief Title: Effect of PEEP on TRJV in Mechanically Intubated Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Iris Mandell, Assistant Professor, Donald and Barbara Zucker School of Medicine at Hofstra/Northwell, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 23-0615
Record Dates: First submitted 2024-01-09; First posted 2024-01-29 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Tricuspid Regurgitation; Mechanical Ventilation Pressure High; Pediatric Respiratory Diseases
Keywords: PEEP; Invasive Mechanical Ventilation; Tricuspid Regurgitant Jet Velocity; Point-of-care-ultrasound
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Participants (Experimental): Application of positive-end-expiratory-pressure on mechanically ventilated patients while performing point-of-care-ultrasound.
  Interventions: Other: Application of positive-end-expiratory pressure

INTERVENTIONS:
Other: Application of positive-end-expiratory pressure — Application of PEEP on mechanically ventilated pediatric patients. Point-of-care-ultrasound performed after each PEEP application.

SUMMARY:
Prospective observational cohort study within the Pediatric Intensive Care Unit (PICU). We will perform point-of-care-ultrasound (POCUS) to quantify tricuspid regurgitant jet velocity (TRJV) on mechanically ventilated (MV) children. Mechanically ventilated (MV) children approaching extubation as per the discretion of the PICU clinical team will undergo a positive end expiratory pressure (PEEP) titration protocol in a safe and timely manner in the PICU. During this PEEP titration, POCUS will be performed by a pediatric intensivist and interpreted by a pediatric cardiologist. Medical demographics will be collected from the electronic medical record and recorded.

DETAILED DESCRIPTION:
New admissions to the PICU will be identified by screening the electronic medical record (EMR) and all intubated patients will be screened and approached for enrollment if they meet inclusion criteria. After informed consent is obtained, subjects will be assigned a unique identifying number. Data will be stored in REDCap. A master link connecting subject POCUS image will be locked in the PI's office.

1. POCUS measurements: POCUS will be performed when a patient is determined to meet extubation readiness criteria as decided by the PICU clinical team. When the patient is on extubation readiness trial (ERT) settings (PEEP baseline), POCUS will be performed to assess TRJV. The PEEP will be increased to PEEP baseline+3 for 15 minutes followed by a repeat POCUS to assess TRJV. The PEEP will then be increased to PEEP baseline+5 (for a max total PEEP of 10mmHg) for 15 minutes followed by a repeat POCUS to assess TRJV. The patients will then be returned to baseline ERT (PEEP baseline) settings prior to the initial POCUS.
2. Interrater reliability will be evaluated amongst trained ultrasound providers by means of performing double scans for 25% of all scans performed. Each subject included in the study will have 3 scans in total (scan at PEEP baseline, scan at PEEP baseline+3, scan at PEEP baseline+5). Since the total number of scans in this study is 90, the number of double scans performed for interrater reliability will be about 22. Each double scan will include an expert ultrasound provider, along with novice ultrasound providers, who will be collecting data for this study. The novice ultrasound provider will participate in a brief informational session of how to obtain and interpret images with the expert provider.
3. Images will be stored in QPATH (our secure ultrasound-image database) and will not have any patient identifiers included. In addition, the attending of record will be contacted to determine if there are any extenuating medical or social circumstances that they believe should preclude the research team from performing the POCUS. If there are, the research team will forgo the POCUS.
4. The POCUS will then be reviewed by a board certified cardiologist and measurements of the TRJV will be obtained. The cardiologist will be blinded to the patient.
5. Information will be obtained from the EMR as outlined in our data collection sheet.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to Cohen Children's Medical Center (CCMC) PICU who are age 3 months - 18 years old who are invasively mechanically ventilated (oral or nasotracheally).
* Patients on or approaching extubation readiness trial.
* Patients with structurally normal heart.
* Patients with normally functioning heart.
* Consent by a legal guardian.

Exclusion Criteria:

* Patients with known air-leak syndrome.
* Patients with history of congenital heart disease (CHD) (pre/post repair).
* Patients with significant cardiac dysfunction and/or on vasoactive medications.
* Patients with history of cardiomyopathy.
* Patients with history of pulmonary hypertension.
* Patients with history of chronic respiratory failure.
* Patients with known mediastinal mass.
* Patients with tracheostomy.

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2023-12-06 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-09-21 (Actual)

PRIMARY OUTCOMES:
Tricuspid Regurgitant Jet Velocity | 30 minutes
  The primary endpoint for the study will be TRJV at baseline PEEP (PEEP baseline) and subsequent PEEP increments (PEEP baseline+3, PEEP baseline+5).

SECONDARY OUTCOMES:
Systolic Blood Pressure | 30 minutes
  mmHg
Diastolic Blood Pressure | 30 minutes
  mmHg
Mean Arterial Pressure | 30 Minutes
  mmHg
Heart Rate | 30 minutes
  BPM (beats per minute)

CONTACTS AND LOCATIONS:
Locations (1):
- Cohen Children's Medical Center, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Artucio H, Hurtado J, Zimet L, de Paula J, Beron M. PEEP-induced tricuspid regurgitation. Intensive Care Med. 1997 Aug;23(8):836-40. doi: 10.1007/s001340050419. PMID 9310800
- [Background] Binder ZW, O'Brien SE, Boyle TP, Cabral HJ, Sekhavat S, Pare JR. Novice Physician Ultrasound Evaluation of Pediatric Tricuspid Regurgitant Jet Velocity. West J Emerg Med. 2020 Jun 24;21(4):1029-1035. doi: 10.5811/westjem.2020.3.45882. PMID 32726279
- [Background] Binder ZW, O'Brien SE, Boyle TP, Cabral HJ, Pare JR. Tricuspid Regurgitant Jet Velocity Point-of-Care Ultrasound Curriculum Development and Validation. POCUS J. 2021 Nov 23;6(2):88-92. doi: 10.24908/pocus.v6i2.15190. PMID 35899222
- [Background] Brower RG, Lanken PN, MacIntyre N, Matthay MA, Morris A, Ancukiewicz M, Schoenfeld D, Thompson BT; National Heart, Lung, and Blood Institute ARDS Clinical Trials Network. Higher versus lower positive end-expiratory pressures in patients with the acute respiratory distress syndrome. N Engl J Med. 2004 Jul 22;351(4):327-36. doi: 10.1056/NEJMoa032193. PMID 15269312
- [Background] Jone PN, Ivy DD. Echocardiography in pediatric pulmonary hypertension. Front Pediatr. 2014 Nov 12;2:124. doi: 10.3389/fped.2014.00124. eCollection 2014. PMID 25429362
- [Background] Jullien T, Valtier B, Hongnat JM, Dubourg O, Bourdarias JP, Jardin F. Incidence of tricuspid regurgitation and vena caval backward flow in mechanically ventilated patients. A color Doppler and contrast echocardiographic study. Chest. 1995 Feb;107(2):488-93. doi: 10.1378/chest.107.2.488. PMID 7842782
- [Background] Khandelwal A, Kapoor I, Mahajan C, Prabhakar H. Effect of Positive End-Expiratory Pressure on Optic Nerve Sheath Diameter in Pediatric Patients with Traumatic Brain Injury. J Pediatr Neurosci. 2018 Apr-Jun;13(2):165-169. doi: 10.4103/jpn.JPN_112_17. PMID 30090129
- [Background] Lai C, Shi R, Beurton A, Moretto F, Ayed S, Fage N, Gavelli F, Pavot A, Dres M, Teboul JL, Monnet X. The increase in cardiac output induced by a decrease in positive end-expiratory pressure reliably detects volume responsiveness: the PEEP-test study. Crit Care. 2023 Apr 9;27(1):136. doi: 10.1186/s13054-023-04424-7. PMID 37031182
- [Background] Persson JN, Kim JS, Good RJ. Diagnostic Utility of Point-of-Care Ultrasound in the Pediatric Cardiac Intensive Care Unit. Curr Treat Options Pediatr. 2022;8(3):151-173. doi: 10.1007/s40746-022-00250-1. Epub 2022 Jul 8. PMID 36277259
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Background] Watkins LA, Dial SP, Koenig SJ, Kurepa DN, Mayo PH. The Utility of Point-of-Care Ultrasound in the Pediatric Intensive Care Unit. J Intensive Care Med. 2022 Aug;37(8):1029-1036. doi: 10.1177/08850666211047824. Epub 2021 Oct 9. PMID 34632837